CLINICAL TRIAL: NCT02586623
Title: RESTORE: A Clinical Study of Patients With Symptomatic Neurogenic Orthostatic Hypotension to Assess Sustained Effects of Droxidopa Therapy
Brief Title: Sustained Effect of Droxidopa in Symptomatic Neurogenic Orthostatic Hypotension
Acronym: RESTORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16306A; NOH402 (Other: NOH402)
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension
Keywords: Parkinson's Disease; Multiple System Atrophy; Pure Autonomic Failure; Primary Autonomic Failure; Dopamine Beta Hydroxylase Deficiency
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Pure Autonomic Failure; dopamine beta hydroxylase deficiency | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Label Period (Experimental): Active droxidopa 100, 200, 300, 400, 500, or 600 mg three times daily (TID) orally. During the Open Label Titration Period, patients will first receive 100 mg TID and their dose will be raised (in 100 mg increments) at subsequent visits until optimal dose is determined. During the Open Label Treatment Period, patients will receive active droxidopa100, 200, 300, 400, 500, or 600 mg three times daily (TID) orally (equal to the patient's individual dose at the end of the Open-Label Titration Period).
  Interventions: Drug: Droxidopa capsules
- Randomized Period (Placebo Comparator): Active droxidopa 100, 200, 300, 400, 500, or 600 mg three times daily (TID) orally (equal to patients individual dose at the end of the Open-Label Period) or matching placebo.
  Interventions: Drug: Droxidopa capsules; Drug: Placebo capsules

INTERVENTIONS:
Drug: Droxidopa capsules — 100, 200 or 300 mg
  Other Names: Northera
Drug: Placebo capsules
  Other Names: Placebo
  Arms: Randomized Period

SUMMARY:
To evaluate the time to treatment intervention in patients with Parkinson's Disease (PD), Multiple System Atrophy (MSA), Pure Autonomic Failure (PAF), Non-Diabetic Autonomic Neuropathy (NDAN) or Dopamine Beta Hydroxylase (DBH) Deficiency who have been previously stabilized with droxidopa therapy for symptoms of neurogenic orthostatic hypotension (NOH) (dizziness, light-headedness, or feelings that they are about to black out)

DETAILED DESCRIPTION:
This is a multi-site, placebo-controlled, double-blind, randomized withdrawal, time to intervention study with a duration of up to 36 weeks, consisting of 5 periods:

Screening Period: up to 4 weeks duration; Open-Label Titration Period (Titration Period): up to 4 weeks duration; Open-Label Treatment Period (Open-Label Period): 12 weeks duration; Double-Blind Treatment Period (Double-Blind Period): 12 weeks duration; Safety Follow-Up Period: 4 weeks duration

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and able to stand (with or without limited assistance)
* Clinical diagnosis of symptomatic orthostatic hypotension associated with Primary Autonomic Failure (PD, MSA or PAF) or NDAN or DBH Deficiency
* Score of at least 4 or greater on Orthostatic Hypotension Symptom Assessment (OHSA) Item #1 (measured at Screening [Visit 1] and the first Titration Visit [Visit 2a] prior to dosing)
* A documented drop of at least 20 millimeters of mercury (mmHg) in SBP, within 3 minutes of standing. This can either be documented in the patient history or assessed during Screening prior to the first Titration Visit (Visit 2a)
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care

Additional inclusion criteria for patients taking prescribed droxidopa prior to study entry:

Patients who are taking prescribed droxidopa therapy are eligible to participate in the study if they meet the other inclusion criteria and also have been on a stable dose of prescribed droxidopa for at least 2 weeks prior to the Screening Visit (Visit 1). In addition, they must meet either of the following at the Screening Visit (Visit 1):

* The patient's Visit 1 OHSA Item #1 score is ≥ 7 AND the prescribed dose is ≤ 300 mg three times daily (TID); OR
* The patient's Visit 1 OHSA Item #1 score is ≤6 AND worsens by ≥ 2 units when retested after washing out of droxidopa for at least 3 days

Exclusion Criteria:

* In the investigator's opinion, the patient is not able to understand or cooperate with study procedures
* Known or suspected alcohol or substance use disorder within the past 12 months (DSM-5 criteria)
* Women who are pregnant or breastfeeding
* Women of childbearing potential (WOCP) who are not using at least one method of contraception with their partner
* Sustained supine hypertension greater than or equal to 180 mmHg systolic or 110 mmHg diastolic. Sustained is defined as the average of 3 observations each at least 10 minutes apart with the patient having been supine and at rest for at least 5 minutes prior to each measurement.
* Untreated closed angle glaucoma
* Diagnosis of hypertension that requires treatment with antihypertensive medications (short-acting antihypertensives to treat nocturnal supine hypertension are allowed in this study)
* Any significant uncontrolled cardiac arrhythmia
* History of myocardial infarction or stroke, within the past 2 years
* Current unstable angina
* Congestive heart failure (NYHA Class 3 or 4)
* Diabetic autonomic neuropathy
* History of cancer within the past 2 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ
* Any major surgical procedure within the past 30 days
* Currently receiving any investigational drug or have received an investigational drug within the past 28 days

Additional protocol defined exclusion criteria do apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (168):
- United States (168):
  - MDFirst Research - Chandler, Chandler, Arizona
  - 21st Century Neurology, Phoenix, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Center For Neurosciences, Tucson, Arizona
  - Movement Disorder Clinic - The University of Arizona, Tucson, Arizona
  - University of Arizona Health Sciences Center, Department Of Neurology, Tucson, Arizona
  - Arkansas Cardiology Clinic, Little Rock, Arkansas
  - East Bay Physicians Medical Group, Berkeley, California
  - Sutter East Bay Medical Foundation, Berkeley, California
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University Of Southern California, Los Angeles, California
  - Parkinson's Institute and Clinical Center, Mountain View, California
  - Diverse Research Solutions, LLC, Oxnard, California
  - Focilmed, Oxnard, California
  - Parkinsons Disease & Movement Disorder of Silicon Valley, Palo Alto, California
  - Neurosearch, Inc. - Pasedena, Pasadena, California
  - Neurosearch, Inc. - Ventura, Pasadena, California
  - SC3 Research Group, Pasadena, California
  - Neurosearch, Inc. - Reseda, Reseda, California
  - Radiological Associates of Sacramento, Sacramento, California
  - Sutter Neuroscience, Sacramento, California
  - The Parkinson's Institute and Clinical Center, Sunnyvale, California
  - Neurosearch Inc. - Torrance, Torrance, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Associated Neurologists, P.C., Danbury, Connecticut
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - Eastern Connecticut Neurology Specialists, LLC, Manchester, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Yale Neurology / Hypertension Program, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Christiana Care Neurology Specialists, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - MedStar Georgetown-MedStar Georgetown Transplant Institute University Hospital (MGUH), Washington D.C., District of Columbia
  - Neurology Offices Of South Florida, Boca Raton, Florida
  - Parkinson's Disease And Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - South Florida Neurology Associates, P.A., Boca Raton, Florida
  - Innovative Research of West Florida, Clearwater, Florida
  - UF Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Galiz Research, Hialeah, Florida
  - SIH Research, Kissimmee, Florida
  - Neurology Associates, Maitland, Florida
  - Future Clinical Research, Miami, Florida
  - Project 4 Research, Miami, Florida
  - Premium Medical Research, Corp, Miami, Florida
  - University Of Miami - Jackson Memorial Hospital, Dept. of Neurology, Miami, Florida
  - Coral Way Research, Miami, Florida
  - Florida Research Center, Miami, Florida
  - Anchor Medical Research, LLC, Miami, Florida
  - Novel Clinical Research Center, LLC, Miami, Florida
  - Pro-Care Research Center, Corporation, Miami Gardens, Florida
  - New Life Medical Research Center, Miami Lakes, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Eminance Medical & Clinical Research, Tampa, Florida
  - University Of South Florida, Tampa, Florida
  - USF Parkinson's & Movement Disorders Center, Tampa, Florida
  - Vero Neurology, Vero Beach, Florida
  - Geodyssey Research, LLC, Vero Beach, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Neurological Center of North Georgia, Gainesville, Georgia
  - The Neurological Center of North Georgia, Gainesville, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Northwestern Medical Group, Chicago, Illinois
  - Cardio Specialists Group, Ltd., Rush University Medical Center, Chicago, Illinois
  - Rush University Medical Center - Department Of Cardiology, Chicago, Illinois
  - Rush University Medical Center, Department of Neurology, Chicago, Illinois
  - NorthShore Neurological Institute, Glenview, Illinois
  - Central Dupage Hospital, Winfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - American Health Network of Indiana, Avon, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Franciscan Physician Network Indiana Heart Physicians, Indianapolis, Indiana
  - Mid America Cardiology - University of Kansas, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana Heart Center, Covington, Louisiana
  - Maine Medical Partners Technology, Scarborough, Maine
  - Mir Neurology, Hagerstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Movement Disorders Clinic, Boston, Massachusetts
  - Movement Disorders Clinic, Boston, Massachusetts
  - Autonomic and Movement Disorders, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital (BWFH) - Brigham & Women's Foot & Ankle Center, Boston, Massachusetts
  - Michigan State University, Department of Neurology, East Lansing, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Nothern Michigan Neurology, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Platte Valley Medical Group, Kearney, Nebraska
  - Methodist Physicians Clinic - Heart Consultants, Omaha, Nebraska
  - MPC Heart Consultants, Omaha, Nebraska
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - JFK Neuroscience Institution, Edison, New Jersey
  - Neuroscience Research Institute, LLC, Toms River, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - David L. Kreitzman MD, PC, Commack, New York
  - Office of David L. Kreitzman, M.D., P.C., Commack, New York
  - Neurology Associates of West Chester, Hawthorne, New York
  - Parker Jewish Institute for Health Care & Rehabilitation, New Hyde Park, New York
  - Weill Cornell Medical College, Dept. of Neurology, New York, New York
  - The Bendheim Parkinson and Movement Disorders Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Project 4 Research, Inc., The Neurological Institute at Columbia University Medical Center, New York, New York
  - The Neurological Institute at Columbia University Medical Center, New York, New York
  - Parker Jewish Institute For Healthcare And Rehabilitation, New York, New York
  - Island Neurological Associates, Plainview, New York
  - Alpha Neurology, Staten Island, New York
  - Helen Hayes Hospital, West Haverstraw, New York
  - UBMD Neurology, Williamsville, New York
  - Peak Clinical Trials, Apex, North Carolina
  - The Neurological Institute, PA, Charlotte, North Carolina
  - Neurosciences Institute, Charlotte, North Carolina
  - Carolinas HealthCare System Neurosciences Institute, Charlotte, North Carolina
  - Insight Neuroscience, LLC, Bellevue, Ohio
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Riverhills Healthcare, Inc., Cincinnati, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Ohio State University, Department of Neurology, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Gardner-McMaster Parkinson Center - The University of Toledo, Toledo, Ohio
  - Medical College of Ohio, Department of Neurology, Toledo, Ohio
  - Baha Abu-Esheh, MD, Ardmore, Oklahoma
  - CardioVoyage, LLC, Ardmore, Oklahoma
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Legacy / Oregon Clinic Neurology, Portland, Oregon
  - The Oregon Clinic, Portland, Oregon
  - St. Luke's Neurology Associates, Bethlehem, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel Neurosciences Institute, Philadelphia, Pennsylvania
  - University of Pennsylvania, Parkinson's Disease & Movement Disorders Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Department of Neurology, Pittsburgh, Pennsylvania
  - Dr. Umer Akbar MD, Office of, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Autonomic Dysfunction Center - Clinical Trials Center, Nashville, Tennessee
  - iMD Medical Center, Carrollton, Texas
  - Sunbeam Clinical Research, Carrollton, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Elite Primary Care, Greenville, Texas
  - Sunbeam Clinical Research, Greenville, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Institute of Cardiology, The Heartbeat Clinic, McKinney, Texas
  - The Heartbeat Clinic, McKinney, Texas
  - Sunbeam Clinical Research, LLC., Prosper, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Christus Research Institute, Tyler, Texas
  - Clear Lake Specialties, Webster, Texas
  - Bateman Home Center, Salt Lake City, Utah
  - Inova Health Systems, Alexandria, Virginia
  - Integrated Neurology Services, PLLC, Falls Church, Virginia
  - Health Research of Hampton Roads-Norfolk, Inc, Norfolk, Virginia
  - Sentara Neurology Specialists, Norfolk, Virginia
  - Henrico Doctors Neurology Associates, LLC, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Northwest Neurology, Premier Clinical Research, Spokane, Washington
  - Premeir Clinical Research, Spokane, Washington
  - Aurora Medical Center, Grafton, Wisconsin
  - Grafton Medical Office, Grafton, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Department of Neurology, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center-Arrhythmia Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hauser RA, Favit A, Hewitt LA, Lindsten A, Gorny S, Kymes S, Isaacson SH. Durability of the Clinical Benefit of Droxidopa for Neurogenic Orthostatic Hypotension During 12 Weeks of Open-Label Treatment. Neurol Ther. 2022 Mar;11(1):459-469. doi: 10.1007/s40120-021-00317-5. Epub 2022 Feb 2. PMID 35107750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 85 sites in the United States. 2 participants were enrolled but excluded from all analysis sets due to incorrect signing of the Informed Consent Form.
Groups:
- Open-Label Droxidopa: Active droxidopa 100, 200, 300, 400, 500, or 600 mg three times daily (TID) orally. During the Open-Label period, participants received 100 mg TID and their dose was raised (in 100 mg TID increments) at subsequent visits until optimal dose was determined. Participants then received active droxidopa 100, 200, 300, 400, 500, or 600 mg TID orally (equal to the participant's individual optimal dose).
- Double-Blind Droxidopa: Active droxidopa 100, 200, 300, 400, 500, or 600 mg TID orally (equal to participant's individual dose at the end of the Open-Label Period)
- Double-Blind Placebo: Matching placebo for droxidopa TID orally
Period: Open-Label (Up to 16 Weeks)
Arm/Group | Open-Label Droxidopa | Double-Blind Droxidopa | Double-Blind Placebo
Started | 453 | 0 | 0
Received at Least 1 Dose of Study Drug | 451 | 0 | 0
Safety Set | 451 | 0 | 0
Completed | 253 | 0 | 0
Not Completed | 200 | 0 | 0
Not completed — Adverse Event | 53 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Non-Compliance | 6 | 0 | 0
Not completed — Physician Decision | 11 | 0 | 0
Not completed — Protocol Violation | 9 | 0 | 0
Not completed — Withdrawal by Subject | 56 | 0 | 0
Not completed — Did not meet Open-label entry criteria | 30 | 0 | 0
Not completed — Did not meet Randomization Criteria | 17 | 0 | 0
Not completed — Incorrect signing of ICF | 2 | 0 | 0
Not completed — Met stopping criteria | 4 | 0 | 0
Not completed — Sponsor request to withdraw | 3 | 0 | 0
Not completed — Discontinued per medical monitor request | 2 | 0 | 0
Not completed — Site closing | 3 | 0 | 0
Period: Double-Blind (Up to 12 Weeks)
Arm/Group | Open-Label Droxidopa | Double-Blind Droxidopa | Double-Blind Placebo
Started | 0 | 127 | 126
Received at Least 1 Dose of Study Drug | 0 | 126 | 126
Full Analysis Set (FAS) | 0 | 126 | 126
Completed | 0 | 78 | 86
Not Completed | 0 | 49 | 40
Not completed — Adverse Event | 0 | 6 | 4
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Non-compliance | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 5
Not completed — Met the need for intervention criteria | 0 | 31 | 27
Not completed — Did not meet randomization criteria | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set (open-label droxidopa) included all participants who received at least one dose of Investigational Medicinal Product (IMP). The Full Analysis Set (double-blind droxidopa, double-blind placebo) included all randomized patients who took at least one dose of IMP in the double-blind period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-Label Droxidopa | Double-Blind Droxidopa | Double-Blind Placebo | Total
Number analyzed (Participants) | 451 | 126 | 126 | 703
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are being reported separately for the open-label and double-blind periods.
  years
    Open-Label Period: number analyzed (Participants) | 451 | 0 | 0 | 451
    Open-Label Period | 66.3 (15.60) |  |  | 66.3 (15.60)
    Double-Blind Period: number analyzed (Participants) | 0 | 126 | 126 | 252
    Double-Blind Period |  | 64.8 (16.10) | 64.6 (15.76) | 64.7 (15.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind periods.
  Participants
    Open-Label Period: number analyzed (Participants) | 451 | 0 | 0 | 451
    Open-Label Period: Female | 196 |  |  | 196
    Open-Label Period: Male | 255 |  |  | 255
    Double-Blind Period: number analyzed (Participants) | 0 | 126 | 126 | 252
    Double-Blind Period: Female |  | 56 | 61 | 117
    Double-Blind Period: Male |  | 70 | 65 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind periods.
  Participants
    Open-Label Period: number analyzed (Participants) | 451 | 0 | 0 | 451
    Open-Label Period: Hispanic or Latino | 86 |  |  | 86
    Open-Label Period: Not Hispanic or Latino | 365 |  |  | 365
    Open-Label Period: Unknown or Not Reported | 0 |  |  | 0
    Double-Blind Period: number analyzed (Participants) | 0 | 126 | 126 | 252
    Double-Blind Period: Hispanic or Latino |  | 32 | 46 | 78
    Double-Blind Period: Not Hispanic or Latino |  | 94 | 80 | 174
    Double-Blind Period: Unknown or Not Reported |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind periods.
  Participants
    Open-Label Period: number analyzed (Participants) | 451 | 0 | 0 | 451
    Open-Label Period: American Indian or Alaska Native | 2 |  |  | 2
    Open-Label Period: Asian | 11 |  |  | 11
    Open-Label Period: Native Hawaiian or Other Pacific Islander | 2 |  |  | 2
    Open-Label Period: Black or African American | 15 |  |  | 15
    Open-Label Period: White | 421 |  |  | 421
    Open-Label Period: More than one race | 0 |  |  | 0
    Open-Label Period: Unknown or Not Reported | 0 |  |  | 0
    Double-Blind Period: number analyzed (Participants) | 0 | 126 | 126 | 252
    Double-Blind Period: American Indian or Alaska Native |  | 0 | 1 | 1
    Double-Blind Period: Asian |  | 1 | 3 | 4
    Double-Blind Period: Native Hawaiian or Other Pacific Islander |  | 2 | 0 | 2
    Double-Blind Period: Black or African American |  | 5 | 4 | 9
    Double-Blind Period: White |  | 118 | 118 | 236
    Double-Blind Period: More than one race |  | 0 | 0 | 0
    Double-Blind Period: Unknown or Not Reported |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time To Intervention
Description: Kaplan-Meier estimates are presented for time to treatment intervention. The estimates represent the quartiles of the survival time, where 50% corresponds to the median time to need for treatment intervention.
  Need for intervention is defined as meeting ANY of the following criteria during the Double-Blind Treatment Period:
  * OHSA Item #1 ≥2 unit worsening from Randomization (Visit 6) AND lack of efficacy as judged by the investigator; OR
  * OHSA Item #1 ≥2 unit worsening from Randomization (Visit 6) at 2 consecutive visits; OR
  * OHSA Item #1 ≥2 unit worsening from Randomization (Visit 6) at the visit before early discontinuation; OR
  * participant stops IMP or withdraws from study for patient-reported lack of efficacy.
Time Frame: Randomization (Day 0) up to Week 12
Population: The Full-analysis Set (FAS) included all randomized participants who took at least one dose of IMP in the Double-Blind Treatment Period.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 126 | 126
Days
  25% | 52.00 [26.00 to 72.00] | 42.00 [27.00 to 86.00]
  50% | NA [NA to NA] — Insufficient number of events occurred to calculate this value | NA [NA to NA] — Insufficient number of events occurred to calculate this value
  75% | NA [NA to NA] — Insufficient number of events occurred to calculate this value | NA [NA to NA] — Insufficient number of events occurred to calculate this value
Statistical Analysis 1: Comparison: Double-Blind Droxidopa vs Double-Blind Placebo; Test type: Superiority; p = 0.803, Log Rank; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.67 to 1.62] — Droxidopa / Placebo

2. Secondary Outcome: Number of Participants Who Needed Intervention During the 12-week Double-Blind Treatment Period
Description: Need for intervention is defined as meeting ANY of the following criteria during the Double-Blind Treatment Period:
  * OHSA Item #1 ≥2 unit worsening from Randomization (Visit 6) AND lack of efficacy as judged by the investigator; OR
  * OHSA Item #1 ≥2 unit worsening from Randomization (Visit 6) at 2 consecutive visits; OR
  * OHSA Item #1 ≥2 unit worsening from Randomization (Visit 6) at the visit before early discontinuation; OR
  * participant stops IMP or withdraws from study for patient-reported lack of efficacy.
Time Frame: Randomization (Day 0) up to Week 12
Population: The FAS included all randomized participants who took at least one dose of IMP in the Double-Blind Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 126 | 126
Participants | 41 | 40

3. Secondary Outcome: Time To All-cause Discontinuation
Description: Kaplan-Meier estimates are presented for time to all-cause discontinuation. The estimates represent the quartiles of the survival time, where 50% corresponds to the median time to discontinuation. Time to all-cause discontinuation was defined as the time from randomization to withdrawal or last contact date.
Time Frame: Randomization (Day 0) up to Week 12
Population: The FAS included all randomized participants who took at least one dose of IMP in the Double-Blind Treatment Period.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 126 | 126
Days
  25% | 42.00 [26.00 to 56.00] | 51.00 [28.00 to NA] — Insufficient number of events occurred to calculate this value
  50% | NA [NA to NA] — Insufficient number of events occurred to calculate this value | NA [NA to NA] — Insufficient number of events occurred to calculate this value
  75% | NA [NA to NA] — Insufficient number of events occurred to calculate this value | NA [NA to NA] — Insufficient number of events occurred to calculate this value

4. Secondary Outcome: Change From Randomization To All Post-randomization Visits in Orthostatic Hypotension Symptom Assessment (OHSA) Item #1 Score
Description: The OHSA scale was designed to rate symptoms occurring specifically as a result of low blood pressure (BP), on average, over the past week using an 11-point scale (0 to 10), with more severe symptoms scoring higher. A score of zero indicates that the symptom was not experienced, and 10 is the worst possible. The scale was used to assess six symptoms: 1) Dizziness, lightheadedness, feeling faint, or feeling like you might black out, 2) problems with vision, 3) weakness, 4) fatigue, 5) trouble concentrating, and 6) head/neck discomfort. Scores for each activity and a composite score for all six activities were tabulated. A mean negative change from baseline means that symptoms have improved. A mean positive change from baseline means that symptoms have gotten worse.
Time Frame: Randomization (Day 0); Weeks 2 to 12
Population: The FAS included all randomized participants who took at least one dose of IMP in the Double-Blind Treatment Period. Here, 'Overall number of subjects analyzed' signifies participants evaluable for this outcome measure and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 121 | 124
Score on a scale
  Week 2 | 0.5 (1.94) | 0.5 (1.91)
  Week 4: number analyzed (Participants) | 106 | 109
  Week 4 | 0.3 (1.83) | 0.3 (1.66)
  Week 6: number analyzed (Participants) | 96 | 98
  Week 6 | 0.3 (1.77) | 0.1 (1.41)
  Week 8: number analyzed (Participants) | 92 | 92
  Week 8 | 0.2 (1.93) | 0.0 (1.50)
  Week 10: number analyzed (Participants) | 82 | 84
  Week 10 | -0.3 (1.62) | -0.5 (1.42)
  Week 12: number analyzed (Participants) | 80 | 88
  Week 12 | 0.1 (1.57) | -0.5 (1.52)

5. Secondary Outcome: Change From Randomization To All Post-randomization Visits in Orthostatic Hypotension Questionnaire (OHQ) Composite Score
Description: The OHQ composite score was a mean of the OHSA composite and the Orthostatic Hypotension Daily Activity Scale (OHDAS) composite scores. The OHDAS was designed as a measure of quality of life. It uses an 11-point scale to assess whether orthostatic hypotension (OH) "interfered" with four types of activities: 1) standing for a short time, 2) standing for a long time, 3) walking for a short time, and 4) walking for a long time. A zero rating means that over the preceding week the activity was performed with no interference and a 10 rating means that orthostatic hypotension completely interfered with the activity. Scores for each activity and a composite score for all four activities were tabulated. A mean negative change from baseline means that symptoms have improved. A mean positive change from baseline means that symptoms have gotten worse.
Time Frame: Randomization (Day 0); Weeks 2 to 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 117 | 122
Score on a scale
  Week 2 | 0.41 (1.673) | 0.40 (1.509)
  Week 4: number analyzed (Participants) | 102 | 107
  Week 4 | 0.21 (1.324) | 0.10 (1.281)
  Week 6: number analyzed (Participants) | 95 | 96
  Week 6 | 0.12 (1.257) | -0.05 (1.236)
  Week 8: number analyzed (Participants) | 89 | 90
  Week 8 | 0.10 (1.472) | -0.25 (1.140)
  Week 10: number analyzed (Participants) | 81 | 82
  Week 10 | -0.19 (1.174) | -0.56 (1.153)
  Week 12: number analyzed (Participants) | 78 | 85
  Week 12 | -0.08 (1.467) | -0.57 (1.163)

6. Secondary Outcome: Clinician-rated Clinical Global Impressions - Severity (CGI-S)
Description: The CGI-S was developed to provide global measures of the severity of a participant's clinical condition during clinical studies. The CGI-S was utilized by both the clinician and the participant to provide an impression of the participant's current state of OH. The severity of the participant's current illness was rated by the clinician on a 7-point scale ranging from 1 (normal, no OH) to 7 (among those patients most extremely ill with OH).
Time Frame: Weeks 2 to 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 118 | 120
Score on a scale
  Week 2 | 3.4 (1.24) | 3.3 (1.22)
  Week 4: number analyzed (Participants) | 106 | 108
  Week 4 | 3.1 (1.26) | 3.3 (1.35)
  Week 6: number analyzed (Participants) | 95 | 95
  Week 6 | 3.2 (1.07) | 3.2 (1.14)
  Week 8: number analyzed (Participants) | 92 | 92
  Week 8 | 3.2 (1.11) | 3.1 (1.24)
  Week 10: number analyzed (Participants) | 81 | 82
  Week 10 | 3.0 (1.15) | 3.0 (1.19)
  Week 12: number analyzed (Participants) | 79 | 88
  Week 12 | 3.0 (1.18) | 2.9 (1.09)

7. Secondary Outcome: Participant-rated CGI-S
Description: The CGI-S was developed to provide global measures of the severity of a participant's clinical condition during clinical studies. The CGI-S was utilized by both the clinician and the participant to provide an impression of the participant's current state of OH. The severity of the participant's current illness was rated by the participant on a 7-point scale ranging from 1 (normal, no OH) to 7 (most extremely ill with OH).
Time Frame: Weeks 2 to 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double-Blind Droxidopa | Double-Blind Placebo
Number analyzed (Participants) | 120 | 123
Score on a scale
  Week 2 | 3.4 (1.31) | 3.2 (1.38)
  Week 4: number analyzed (Participants) | 105 | 109
  Week 4 | 3.2 (1.27) | 3.3 (1.33)
  Week 6: number analyzed (Participants) | 96 | 98
  Week 6 | 3.2 (1.17) | 3.1 (1.21)
  Week 8: number analyzed (Participants) | 92 | 92
  Week 8 | 3.2 (1.22) | 3.1 (1.27)
  Week 10: number analyzed (Participants) | 82 | 83
  Week 10 | 3.1 (1.18) | 3.0 (1.26)
  Week 12: number analyzed (Participants) | 80 | 88
  Week 12 | 3.1 (1.29) | 2.8 (1.19)

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose (Up to approximately 8 months)
Arm/Group | Open-Label Droxidopa | Double-Blind Droxidopa | Double-Blind Placebo
All-Cause Mortality (participants affected / at risk) | 6/451 | 1/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 45/451 | 3/126 | 8/126
Other Adverse Events (participants affected / at risk) | 192/451 | 32/126 | 22/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Droxidopa (N=451) | Double-Blind Droxidopa (N=126) | Double-Blind Placebo (N=126)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (5) | 1 (1) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Droxidopa (N=451) | Double-Blind Droxidopa (N=126) | Double-Blind Placebo (N=126)
Nausea (Gastrointestinal disorders) | 43 (54) | 1 (1) | 1 (1)
Fatigue (General disorders) | 24 (27) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 26 (30) | 10 (11) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 49 (83) | 8 (10) | 5 (9)
Dizziness (Nervous system disorders) | 39 (49) | 7 (8) | 5 (7)
Headache (Nervous system disorders) | 69 (90) | 4 (4) | 7 (8)
Hypertension (Vascular disorders) | 24 (27) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT02586623/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02586623/SAP_001.pdf